CLINICAL TRIAL: NCT01347164
Title: Development and Testing of HIV Prevention Interventions Targeting Black MSM/W
Brief Title: Evaluation of a New HIV Prevention Intervention for Black Bisexually-active Men
Acronym: RISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health Management Corporation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5UR6PS001099 (NIH)
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Bisexually-active Men; at Risk for HIV
Keywords: bisexual; HIV prevention
MeSH Terms: conditions — Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Life coaching sessions (Experimental): 6 2-hour counseling session with trained therapist/counselor. The sessions deal with coping and stress reduction as well as sexual health.
  Interventions: Behavioral: RISE life coaching intervention
- HIV counseling session (Active Comparator): One 60-minute counseling session, based on standard HIV counseling content.
  Interventions: Behavioral: HIV Counseling

INTERVENTIONS:
Behavioral: RISE life coaching intervention — 6 2-hour sessions
  Arms: Life coaching sessions
Behavioral: HIV Counseling — Standard one-hour HIV counseling session
  Arms: HIV counseling session

SUMMARY:
Black men who have sex with men (MSM) have the highest rates of HIV infection in the United States and represent a population in need of new HIV prevention interventions. Although 20 to 40% of Black MSM are estimated to have female partners, no interventions tailored to the needs of Black MSM/W have been developed and rigorously evaluated. This project will develop, implement, and evaluate an individual-level intervention (ILI), titled "RISE", that will assist Black MSM/W to reduce their risk for acquiring and transmitting HIV infection. This intervention will address the effect of individual level factors, interpersonal relationships including sexual, peer and family relationships, and socio-cultural influences on the sexual risk behaviors of MSM/W. The intervention will consist of six counseling sessions held between a trained counselor and participant, and will be guided by three theoretical perspectives: an ecological perspective of behavior, stress and coping theory, and social cognitive theory. The COLOURS Organization, the sole agency in Philadelphia dedicated to exclusively serving the Black LGBT community, will be a key collaborator in the development and implementation of the intervention. The evaluation design utilizes a randomized controlled trial to test the effectiveness of the proposed intervention. Chain referral, based on principles of respondent-driven sampling, will be used to recruit 250 HIV-positive and HIV-negative Black bisexually-active men into this study.

The specific aims of this research are to:

* develop a new theoretically-based individual-level HIV prevention intervention culturally tailored to the needs of HIV-positive and HIV-negative Black MSM/W;
* evaluate the intervention with a randomized control group design, using RDS to recruit 250 Black MSM/W who do not inject drugs and who report recent unprotected sex;
* assess the efficacy of the intervention and test the intervention model through the collection of behavioral risk assessments and HIV and STD testing at three time points: baseline, immediately post-intervention and three-months post-intervention;
* examine and describe individual factors, interpersonal relationships and network factors, and socio-cultural factors that may affect risk behaviors for HIV infection and transmission among Black MSM/W;
* develop recommendations for recruiting Black bisexually-active men and providing them with targeted HIV prevention interventions.

Evaluation data collection will be conducted using ACASI. Data analysis will include Repeated Measures ANOVA to make assessments of changes over time and intervention dose effects and structural equation modeling to assess causal associations between factors in the conceptual model. This proposed study has significance for increasing our understanding various types of factors that may affect sexual risk behaviors of Black MSM/W as well as potentially providing an important new tool for HIV prevention specifically targeting the needs and risk behaviors of Black MSM/W.

ELIGIBILITY:
Inclusion Criteria:

* male and female sex partners past 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
increased condom use | at follow-up 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Lauby, PhD, Principal Investigator — Public Health Management Corporation
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States